CLINICAL TRIAL: NCT07104591
Title: Expanded Access Use of Multivirus-Specific Cytotoxic T-Lymphocytes for Pediatric Patients With EBV, CMV, Adenovirus, or BK Virus Infections Post Allogeneic Stem Cell Transplant
Brief Title: TETRAVI Expanded Access Program
Status: Available | Type: Expanded Access
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: H-44843 TETRAVI EAP
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Epstein-Barr Virus Infection; Cytomegalovirus Infections; Adenovirus Infection; BK Virus Infection; JC Virus Infection; Viral Infections Post-Transplant; Post-Allogeneic Stem Cell Transplant Complications
MeSH Terms: conditions — Epstein-Barr Virus Infections; Cytomegalovirus Infections; Adenoviridae Infections

STUDY DESIGN:
Expanded Access Types: Individual, Treatment

INTERVENTIONS:
Biological: HLA-matched VSTs (Multivirus-specific Cytotoxic T Lymphocytes) — Banked, partially HLA-matched virus-specific T cells (VSTs) directed against EBV, CMV, adenovirus, and BK virus.

SUMMARY:
This Expanded Access Program (EAP) allows qualified physicians within Texas to obtain access to multivirus-specific cytotoxic T lymphocytes (VSTs) developed under Baylor College of Medicine's TETRAVI program (NCT04013802) for the treatment of persistent or recurrent infections with EBV, CMV, adenovirus, or BK virus in pediatric patients being treated in Texas who have received allogeneic stem cell transplants and have no other suitable therapeutic options.

DETAILED DESCRIPTION:
This EAP is limited to pediatric patients being treated in the State of Texas. In this program, Baylor College of Medicine's Center for Cell and Gene Therapy (CAGT) will provide applicable physicians with copies of a template protocol and consent form, allowing each site to establish its own single-patient expanded access protocol. Baylor will also issue a Letter of Authorization (LOA) to cross-reference its own IND. This LOA will accompany the local site's submission to the FDA. The VSTs will be provided to eligible patients through this mechanism upon IRB and FDA approval of the treating site's individual patient protocol.

The aim is to enable access to off-the-shelf partially HLA-matched virus-specific T cells for pediatric patients located in Texas (USA) with limited treatment options due to persistent or resistant viral infections post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients <18 years of age.
* Patients who have undergone myeloablative or non-myeloablative allogeneic HSCT or CAR T therapy in the Sate of Texas (USA).
* Have persistent, increasing, or recurrent infections with EBV, CMV, adenovirus, or BK virus despite standard treatment.
* Treating physician must be based in Texas.
* Must obtain IRB approval and submit a protocol to FDA with Letter of Authorization from Baylor.

Exclusion Criteria:

* Patients with active uncontrolled infections unrelated to the viruses mentioned.
* Use of certain immunosuppressive agents within 28 days.
* Serious uncontrolled medical conditions or relapse of underlying disease.

Max Age: 17 Years | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: John Craddock, MD, Study Chair — Baylor College of Medicine